CLINICAL TRIAL: NCT03006705
Title: A Multicenter, Double-blind, Randomized Study in Patients With Gastric Cancer Undergoing Postoperative Adjuvant Chemotherapy
Brief Title: Study of Adjuvant ONO-4538 With Resected Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ONO-4538-38
Record Dates: First submitted 2016-12-27; First posted 2016-12-30 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Gastric Cancer
Keywords: ONO-4538,BMS-936558,Nivolumab,gastric,adjuvant,S-1,CapeOX
MeSH Terms: conditions — Stomach Neoplasms | interventions — Nivolumab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nivolumab group (Experimental): Nivolumab: 360 mg solution intravenously for 30 min in every 3 weeks (maximum 1 year).
  Chemotherapy: S-1 Therapy or CapeOX Therapy is determined by the investigator.
  S-1 therapy(maximum 1 year):
  Tegafur-gimeracil-oteracil potassium combination drug 40 - 60 mg bid orally in 28 days, followed by 14 days off
  CapeOX Therapy(maximum 6 months):
  Oxaliplatin 130 mg/m2 (body surface area) solution intravenously for 2 hours once-daily, followed by 20 days off.
  Capecitabine 1000 mg2 (body surface area) bid orally in 14 days, followed by 7 days off.
  Interventions: Drug: Nivolumab; Drug: Tegafur-gimeracil-oteracil potassium; Drug: Oxaliplatin; Drug: Capecitabine
- Placebo group (Placebo Comparator): Placebo: Placebo solution intravenously for 30 min in every 3 weeks (maximum 1 year).
  Chemotherapy: S-1 Therapy or CapeOX Therapy is determined by the investigator.
  S-1 therapy(maximum 1 year):
  Tegafur-gimeracil-oteracil potassium combination drug 40 - 60 mg bid orally in 28 days, followed by 14 days off
  CapeOX Therapy(maximum 6 months):
  Oxaliplatin 130 mg/m2 (body surface area) solution intravenously for 2 hours once-daily, followed by 20 days off.
  Capecitabine 1000 mg2 (body surface area) bid orally in 14 days, followed by 7 days off.
  Interventions: Drug: Tegafur-gimeracil-oteracil potassium; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Placebo

INTERVENTIONS:
Drug: Nivolumab — Nivolumab: 360 mg solution intravenously for 30 min in every 3 weeks (maximum 1 year).
  Other Names: BMS-936558; ONO-4538; MDX-1106
  Arms: Nivolumab group
Drug: Tegafur-gimeracil-oteracil potassium — Tegafur-gimeracil-oteracil potassium combination drug 40 - 60 mg bid orally in 28 days, followed by 14 days off
Drug: Oxaliplatin — Oxaliplatin 130 mg/m2 (body surface area) solution intravenously for 2 hours once-daily, followed by 20 days off.
Drug: Capecitabine — Capecitabine 1000 mg2 (body surface area) bid orally in 14 days, followed by 7 days off.
Drug: Placebo — Placebo: 360 mg solution intravenously for 30 min in every 3 weeks (maximum 1 year).
  Arms: Placebo group

SUMMARY:
The purpose of study is to evaluate the efficacy and safety of postoperative adjuvant chemotherapy with Nivolumab in combination with tegafur-gimeracil-oteracil potassium (S-1 therapy) or capecitabine + oxaliplatin (CapeOX therapy), in comparison with placebo in combination with S-1 therapy or CapeOX therapy, in pStage III gastric cancer (including esophagogastric junction cancer) after D2 or more extensive lymph node dissection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed adenocarcinoma of the stomach
* Patients without a remnant cancer (R0) who have undergone gastrectomy
* Gastric carcinoma according to the stage classification of AJCC/UICC TNM Classification, 7th Edition on the basis of overall postoperative findings
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 or 1

Exclusion Criteria:

* Patients who have received non-surgical treatment (e.g., radiotherapy, chemotherapy, hormone therapy) for gastric cancer
* Multiple primary cancers
* A current or past history of severe hypersensitivity to any other antibody products
* Any concurrent autoimmune disease or past history of chronic or recurrent autoimmune disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) | 5 years

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
3-year OS rate | 3 years
5-year OS rate | 5 years
3-year RFS rate | 3 years
5-year RFS rate | 5 years
Safety will be analyzed through the incidence of adverse events, serious adverse events | Up to 28 days from last dose
Safety will be analyzed through the incidence of laboratory abnormalities | Up to 28 days from last dose

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (108):
- China (21):
  - Anhui Province Clinical Site, Anhui Province
  - Beijing Clinical Site1, Beijing
  - Beijing Clinical Site2, Beijing
  - Cuangdong Province Clinical Site, Cuangdong Province
  - Guangdong Province Clinical Site1, Guangdong Province
  - Guangdong Province Clinical Site2, Guangdong Province
  - Henan Province Clinical Site1, Henan Province
  - Henan Province Clinical Site2, Henan Province
  - Jiangsu Province Clinical Site1, Jiangsu Province
  - Jiangsu Province Clinical Site3, Jiangsu Province
  - Jiangsu Province Clinical Site4, Jiangsu Province
  - Jiangsu Province Clinical Site5, Jiangsu Province
  - Jiangsu Province Clinical Site6, Jiangsu Province
  - Jiangxi Province Clinical Site2, Jiangxi Province
  - Jilin Province Clinical Site, Jilin Province
  - Liaoning Province Clinical Site, Liaoning Province
  - Shanxi Province Clinical Site, Shanxi Province
  - Tianjin Clinical Site1, Tianjin
  - Tianjin Clinical Site2, Tianjin
  - Zhejiang Province Clinical Site, Zhejiang Province
  - Zhengjiang Province Clinical Site, Zhengjiang Province
- Japan (55):
  - Aichi Clinical Site1, Nagoya, Aichi-ken
  - Aichi Clinical Site2, Nagoya, Aichi-ken
  - Chiba Clinical Site, Kamogawa, Chiba
  - Ehime Clinical Site, Matsuyama, Ehime
  - Ehime Clinicla Site, Matsuyama, Ehime
  - Gifu Clinical Site, Ōgaki, Gifu
  - Gunma Clinical Site, Ōta, Gunma
  - Gunma Clinical Site, Takasaki, Gunma
  - Hiroshima Clinical Site, Fukuyama, Hiroshima
  - Hokkaido Clinical Site 3, Hakodate, Hokkaido
  - Hokkaido Clinical Site 1, Sapporo, Hokkaido
  - Hokkaido Clinical Site2, Sapporo, Hokkaido
  - Hyogo Clinical Site, Akashi, Hyōgo
  - Hyogo Clinical Site, Amagasaki, Hyōgo
  - Hyogo Clinical Site, Nishinomiya, Hyōgo
  - Ishikawa Clinical Site, Kanazawa, Ishikawa-ken
  - Iwate Clinical Site, Morioka, Iwate
  - Kanagawa Clinical Site, Sagamihara, Kanagawa
  - Kanagawa Clinical Site, Yokohama, Kanagawa
  - Miyagi Clinical Site, Ōsaki, Miyagi
  - Nagano Clinical Site, Saku, Nagano
  - Okayama Clinical Site, Kurashiki, Okayama-ken
  - Osaka Clinical Site, Hirakata, Osaka
  - Osaka Clinical Site, Ōsaka-sayama, Osaka
  - Osaka Clinical Site, Sakai, Osaka
  - Osaka Clinical Site, Suita, Osaka
  - Osaka Clinical Site, Takatsuki, Osaka
  - Osaka Clinical Site, Toyonaka, Osaka
  - Saitama Clinical Site, Hidaka, Saitama
  - Saitama Clinical Site, Kitaadachi-gun, Saitama
  - Shizuoka Clinical Site, Sunto-gun, Shizuoka
  - Tochigi Clinical Site, Shimotsuke, Tochigi
  - Tokyo Clinical Site, Bunkyo-ku, Tokyo
  - Tokyo Clinical Site, Chuo-ku, Tokyo
  - Tokyo Clinical Site, Koto-ku, Tokyo
  - Tokyo Clinical Site, Shinjuku-ku, Tokyo
  - Chiba Clinical Site, Chiba
  - Fukuoka Clinical Site 1, Fukuoka
  - Fukuoka Clinical Site 2, Fukuoka
  - Gifu Clinical Site, Gifu
  - Hiroshima Clinical Site1, Hiroshima
  - Hiroshima Clinical Site2, Hiroshima
  - Hiroshima Clinical Site3, Hiroshima
  - Kochi Clinical Site, Kochi
  - Kumamoto Clinical Site, Kumamoto
  - Kyoto Clinical Site, Kyoto
  - Niigata Clinical Site, Niigata
  - Osaka Clinical Site1, Osaka
  - Osaka Clinical Site2, Osaka
  - Osaka Clinical Site3, Osaka
  - Osaka Clinical Site4, Osaka
  - Shizuoka Clinical Site, Shizuoka
  - Toyama Clinical Site, Toyama
  - Wakayama Clinical Site, Wakayama
  - Yamagata Clinical Site, Yamagata
- South Korea (24):
  - Busan Clinical Site1, Busan
  - Busan Clinical Site2, Busan
  - Busan Clinical Site3, Busan
  - Daegu Clinical Site1, Daegu
  - Daegu Clinical Site2, Daegu
  - Daegu Clinical Site3, Daegu
  - Daejeon Clinical Site 1, Daejeon
  - Daejeon Clinical Site 2, Daejeon
  - Gwangju Clinical Site, Gwangju
  - Gyeonggi-do Clinical Site1, Gyeonggi-do
  - Gyeonggi-do Clinical Site2, Gyeonggi-do
  - Gyeonggi-do Clinical Site3, Gyeonggi-do
  - Gyeonggi-do Clinical Site4, Gyeonggi-do
  - Gyeonggi-do Clinical Site5, Gyeonggi-do
  - Jeollabuk-do Clinical Site, Jeollabuk-do
  - Seoul Clinical Site 8, Seoul
  - Seoul Clinical Site 9, Seoul
  - Seoul Clinical Site1, Seoul
  - Seoul Clinical Site2, Seoul
  - Seoul Clinical Site3, Seoul
  - Seoul Clinical Site4, Seoul
  - Seoul Clinical Site5, Seoul
  - Seoul Clinical Site6, Seoul
  - Seoul Clinical Site7, Seoul
- Taiwan (8):
  - Kaohsiung Clinical Site2, Kaohsiung City
  - Kaohsiung Clinical Site, Kaohsiung City
  - New Taipei Clinical Site, New Taipei City
  - Taichung Clinical Site, Taichung
  - Tainan Clinical Site2, Tainan
  - Tainan Clinical Site, Tainan
  - Taipei Clinical Site1, Taipei
  - Taipei Clinical Site2, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kang YK, Terashima M, Kim YW, Boku N, Chung HC, Chen JS, Ji J, Yeh TS, Chen LT, Ryu MH, Kim JG, Omori T, Rha SY, Kim TY, Ryu KW, Sakuramoto S, Nishida Y, Fukushima N, Yamada T, Bai LY, Hirashima Y, Hagihara S, Nakada T, Sasako M. Adjuvant nivolumab plus chemotherapy versus placebo plus chemotherapy for stage III gastric or gastro-oesophageal junction cancer after gastrectomy with D2 or more extensive lymph-node dissection (ATTRACTION-5): a randomised, multicentre, double-blind, placebo-controlled, phase 3 trial. Lancet Gastroenterol Hepatol. 2024 Aug;9(8):705-717. doi: 10.1016/S2468-1253(24)00156-0. Epub 2024 Jun 18. PMID 38906161
- [Derived] Chang X, Ge X, Zhang Y, Xue X. The current management and biomarkers of immunotherapy in advanced gastric cancer. Medicine (Baltimore). 2022 May 27;101(21):e29304. doi: 10.1097/MD.0000000000029304. PMID 35623069